CLINICAL TRIAL: NCT04097327
Title: Effect of Ectoin Dermatitis Cream 7% (EHK02) on Skin Hydration and Skin Barrier Function in Patients With Atopic Dermatitis: a Prospective, Clinical Study
Brief Title: Effect of Ectoin Dermatitis Cream 7% on Skin Hydration and Skin Barrier Function
Status: Completed | Type: Observational
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Other Study IDs: btph-043-2019_EHK02
Record Dates: First submitted 2019-09-17; First posted 2019-09-20 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Atopic Dermatitis Eczema
Keywords: Ectoin; Ectoin Dermatitis Cream; Atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ectoin Dermatitis Cream 7% (EHK02) — Application of Ectoin Dermatitis Cream in accordance with the instructions for use

SUMMARY:
The aim of this prospective, uncontrolled clinical study is to evaluate the clinical effect of Ectoin® Dermatitis Cream-EHK02 on skin hydration and transepidermal water loss (TEWL) in subjects with atopic dermatitis after single and multiple applications. Furthermore, data concerning the subjective impression of the study preparation should be collected.

DETAILED DESCRIPTION:
The principle mode of Ectoin is based on the physical interaction of this compatible solute with water. Ectoin® Dermatitis Cream 7% (EHK02) is able to build an Ectoin® Hydro Complex on the skin providing an effective protection against external stress factors, stabilizing the skin barrier and moisturizing the dry skin. In former studies, it has been shown that it can be used for the symptomatic treatment of atopic dermatitis. This study should confirm the efficacy and safety of EHK02.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent form to participate in the study
* Female or male individual between 18 and 65 years in good general health
* Diagnosed atopic dermatitis for ≥ 6 months, in asymptomatic stage (asymptomatic stage means without flare up at the beginning of the study)
* Willingness of the participants to actively participate in the study and to come to the scheduled visits
* Willingness of the participants to discontinue the application of EHK02 in the test area throughout the course of the study

Exclusion Criteria:

* Patient has a skin disease that in the investigator's opinion may interfere with the conduct of the study or the evaluation of the results
* Patient is self-reported to be pregnant, nursing or planning pregnancy during the clinical investigation
* Presence of any disease and/or condition and/or history of diseases and/or conditions that according to the investigator may interfere with the conduct of the investigation or the evaluation of the results (such as abnormal laboratory values, chronic inflammatory diseases, immunosuppressive diseases, autoimmune diseases, malignancies, liver or kidney diseases, severe infectious diseases, systemic diseases)
* Patient has a known allergy against any ingredient of the test products
* Patient is known to have had a substance abuse (drug or alcohol) problem within the previous 12 months
* Patient participates in another clinical trial or has participated in another clinical trial within the last 30 days prior to the first day of investigation
* Patient is involved in the organization of the clinical investigation
* Subjects receiving the following topical or systemic treatments: Glucocorticoids and / or anti-histamines during the previous week and during the study, Cough suppressants and/or corticoids during the previous 4 weeks,Retinoids and/or immunosuppressants during the previous 6 months
* Use of skin care products, dermatological therapeutics, shower oils or solarium visits on the test area 7 days prior to the study and during the study
* Swimming or sauna 24 hours prior to the study and during the study
* Hair removal on the tested areas within the study period and within 3 days prior to the study
* Participation in suction blister and UV studies on the tested areas during the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with atopic dermatitis without flare up (in eczema free interval).
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean corneometer measurement 8 hours after treatment | baseline (pretreatment), 8 hours after first application (post treatment)
  Corneometer is a non-invasive instrument that measures barrier function of the skin surface. Change of skin hydration will be assessed comparing values before (initial condition-pretreatment) and after single application. The electrical capacitance of the skin surface will be expressed digitally in arbitrary units. Three measurements will be performed on each test area and the mean will be used to define the skin barrier function of the stratum corneum.
Change from baseline in mean tewameter measurement 8 hours after treatment | baseline (pretreatment), 8 hours after first application (post treatment)
  Transepidermal water loss (TEWL) is affected by environmental factors as humidity, temperature, the time of year (seasonal variation) and the moisture content of the skin (hydration level). Tewameter is a non-invasive instrument that measures skin hydration. Change of skin hydration will be assessed comparing values before (initial condition-pretreatment) and after single application. The TEWL measurement will be measured three times and the mean than will be used to define skin hydration of the stratum corneum. The hydration of the skin surface will be expressed in g/hm².

SECONDARY OUTCOMES:
Change in skin hydration over time (1, 8, and 24 hours) after single application compared to initial condition (pretreatment). | baseline (pretreatment), 1 hour, 8 hours and 24 hours after first application (post treatment).
  Skin hydration will be measured with a Tewameter. Physicians will measure values before (pretreatment), and after 1, 8 and 24 hours (post application).
Change in skin barrier function over time (1, 8, and 24 h) after single application compared to initial condition (pretreatment). | baseline (pretreatment), 1 hour, 8 hours and 24 hours after first application (post treatment).
  Skin barrier function will be measured with a Corneometer. Physicians will measure values before (pretreatment), and after 1, 8 and 24 hours (post application).
Change from baseline (initial condition) in mean Tewameter measurement 7 days after treatment. | baseline and 7 days after treatment
  Skin hydration will be measured with a Tewameter. Physicians will measure values before (pretreatment), and 7 days after multiple applications.
Change from baseline (initial condition) in mean Corneometer measurement 7 days after treatment. | baseline and 7 days after treatment
  Skin barrier function will be measured with a Corneometer. Physicians will measure values before (pretreatment), and 7 days after multiple applications.

CONTACTS AND LOCATIONS:
Locations (1):
- Centroderm GmbH, Wuppertal, Deutschland, Germany